CLINICAL TRIAL: NCT02912390
Title: Cerclage for Ultrasound-Diagnosed Short Cervix in Twins: A Randomized Controlled Trial
Brief Title: Cerclage for Short Cervix in Twins
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: On Internal Hold
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Laura Vricella, MD, Assistant Professor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 27073a; Cerclage in Twins (Other: Saint Louis University Institutional Review Board)
Record Dates: First submitted 2016-08-02; First posted 2016-09-23 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Short Cervix, Twins
MeSH Terms: interventions — Cerclage, Cervical; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cerclage (Active Comparator): - Macdonald cerclage placed in standard fashion
  Interventions: Procedure: Cerclage
- Expectant management (Active Comparator): - Patient is placed on activity restrictions
  Interventions: Other: Expectant management

INTERVENTIONS:
Procedure: Cerclage — Macdonald cerclage placed in standard fashion
  Arms: Cerclage
Other: Expectant management — placed on activity restrictions: no heavy lifting, frequent reclining, and pelvic rest.
  Arms: Expectant management

SUMMARY:
Through cervical length measurement in uncomplicated twin gestations, women with cervical length ≤ 25 mm will be approached for randomization to cerclage placement or expectant management with activity restriction and treatment of preterm labor

DETAILED DESCRIPTION:
Pregnant women with twin gestations are screened for short cervix with transvaginal cervical length measurements as part of routine care at St. Mary's Health Center (SMHC) and Saint Louis University's (SLUCare) Physician Group. (Transvaginal cervical length measurement every 2 weeks from 16weeks/0days-23weeks/6days weeks, per hospital practice) Women pregnant with twin gestations at SMHC who meet study criteria will undergo transvaginal length screening between 16 and 24 weeks gestation. Those women with transvaginal cervical length measurements at or below 25 mm will be approached for study participation.

If a patient agrees to participate in the trial, they will be randomized in 1:1 fashion to cerclage vs. expectant management.

Participants found to have a vaginal infection by cultures performed at randomization will be treated with appropriate antibiotics per usual institutional practices

Cerclage arm:

- Macdonald cerclage placed in standard fashion: mersilene suture preferred for standardization

Expectant management arm:

- Patient is placed on activity restrictions: no heavy lifting, frequent reclining, and pelvic rest.

If a participant does not consent to participate in the trial, permission to collect their outcome information in an observational manner will be requested.

The neonatal medical record will be reviewed for outcome data on twins, weights, complications, neonatal intensive care unit (NICU) stay, to 28 day after discharge.

ELIGIBILITY:
Inclusion Criteria:

* at least 14 years of age, but less than 55 yrs of age
* must be able to read and write English
* must be able to give informed consent.
* Twin pregnancy

Exclusion Criteria:

* Women with a serious physical or mental illness or condition that would substantially interfere with participation in the study
* membrane prolapse beyond the external cervical os,
* major fetal anomaly in either twins will be excluded from randomization.

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2017-01-12; Primary Completion 2018-03 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
cervical length ≤ 25 mm. | 1 year
  To determine whether cerclage placement in women with twin gestation and cervical length ≤ 25 mm results in pregnancy prolongation.

SECONDARY OUTCOMES:
cervical length ≤ 15 mm. | 1 year
  To perform a planned subgroup analysis with adequate power to determine whether cerclage placement results in pregnancy prolongation in twins gestations with cervical length ≤ 15 mm.

OTHER OUTCOMES:
cervical and vaginal microbiomes | 1 year
  To assess the cervical and vaginal microbiomes as well as presence of vaginal infections to determine potential predictors for spontaneous preterm birth in twin gestations with short cervix

CONTACTS AND LOCATIONS:
Overall Officials: Laura Vricella, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No